CLINICAL TRIAL: NCT04599517
Title: The Most Frequently Preferred Surgical Method In The Treatment Of Sacrococcygeal Pilonidal Disease; Multicenter Cohort Study
Brief Title: The Most Frequently Preferred Surgical Method In The Treatment Of Sacrococcygeal Pilonidal Disease
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, prinicipal investigator, Konya Meram State Hospital
Other Study IDs: HSU Konya HPRC General Surgery
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Pilonidal Sinus
Keywords: pilonidal; surgery; healing
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is no consensus on which procedure is the ideal surgical method in the treatment of sacrococcygeal pilonidal disease (SPD). The study aimed to retrospectively screen the cases that had undergone surgical treatment for SPD in the last 15 years in four different tertiary Stage hospitals and analyze the most frequently used surgical treatment method and its results.

DETAILED DESCRIPTION:
The researchers in our study will retrospectively scan the records of patients who have been operated on for SPD in the last 15 years at Health Sciences University Konya Health Practice and Research Center, Selçuk University Medical Faculty Hospital, Necmettin Erbakan University Medical Faculty Hospital, and Başkent University Medical Faculty Hospital General Surgery Clinics.

Demographic characteristics of the patients, type of anesthesia, duration of operation, duration of hospitalization, time to return to work or school, final healing time, follow-up time, and recurrence information will be transferred to the SPSS statistics program analyzed.

The researchers could not find any articles in the literature on the subject. Therefore, this study will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 14-80 who underwent surgery for pilonidal sinus

Exclusion Criteria:

* unregulated diabetes mellitus
* collagen tissue disease
* decompensated cardiovascular disease
* cases with missing follow-up information

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients aged 14-80 years who underwent surgery for pilonidal sinus constitute the study population.
Sampling Method: Non-Probability Sample
Enrollment: 6748 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Type of surgery method | 15 day
  The ratio of each type of surgery to the study population
duration of surgery | 15 day
  The average operation time of the determined types of surgery will be determined.
hospitalization time | 15 day
  The average hospitalization time of the determined types of surgery will be determined.
Type of anesthesia | 15 day
  the ratio of anesthesia methods to the study population
day time return to work | 15 days
  return to work time will be found as average days for specified surgery types.
complete healing time | 15 days
  Complete healing time will be found as average days for specified surgery types
recurrence | 15 days
  recurrence rate in the study population

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plans to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Johnson EK, Vogel JD, Cowan ML, Feingold DL, Steele SR; Clinical Practice Guidelines Committee of the American Society of Colon and Rectal Surgeons. The American Society of Colon and Rectal Surgeons' Clinical Practice Guidelines for the Management of Pilonidal Disease. Dis Colon Rectum. 2019 Feb;62(2):146-157. doi: 10.1097/DCR.0000000000001237. No abstract available. PMID 30640830
- [Background] Hull TL, Wu J. Pilonidal disease. Surg Clin North Am. 2002 Dec;82(6):1169-85. doi: 10.1016/s0039-6109(02)00062-2. PMID 12516846
- [Background] Stauffer VK, Luedi MM, Kauf P, Schmid M, Diekmann M, Wieferich K, Schnuriger B, Doll D. Common surgical procedures in pilonidal sinus disease: A meta-analysis, merged data analysis, and comprehensive study on recurrence. Sci Rep. 2018 Feb 15;8(1):3058. doi: 10.1038/s41598-018-20143-4. PMID 29449548